CLINICAL TRIAL: NCT03605888
Title: Koa Family: A Study of Improving Diet, Physical Activity, Weight, and Well-being Among Low-income Mothers in California
Brief Title: Koa Family: California's Obesity Prevention Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Department of Health Services (Other); United States Department of Agriculture (USDA) (U.S. Federal Agency); California Department of Social Services (Other Government); CAL FIRE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1229056; 2017-088 (Other: The Committee for the Protection of Human Subjects)
Record Dates: First submitted 2018-07-17; First posted 2018-07-30 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Weight Loss; Diet Habit; Physical Activity; Overweight and Obesity
Keywords: Nutrition
MeSH Terms: conditions — Weight Loss; Feeding Behavior; Motor Activity; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RCT Intervention (Experimental): Overweight or obese (BMI ≥ 25 kg/m2) participants randomized to the Koa Family. intervention
  Interventions: Behavioral: Koa Family
- RCT Control (No Intervention): Overweight or obese (BMI ≥ 25 kg/m2) participants randomized to the control group.
- Exploratory (Other): Normal-weight mothers (BMI 18.5-24.9 kg/m2) assigned to the Koa Family intervention.
  Interventions: Behavioral: Koa Family

INTERVENTIONS:
Behavioral: Koa Family — Koa Family is a 6-month program consisting of a whole-person lifestyle program (WPLP) combined with text messaging and social media support and a neighborhood tree planting campaign. The WPLP will bring groups of 8 to 10 mothers living in the same community together for 22 weekly 90-minute support sessions. Each session will cover a topic on whole-person living, including healthy eating, physical activity, stress reduction, coping, and well-being. Participants will receive brief text messages on their cell phones to encourage healthy lifestyle choices. Participants also will be invited to join a "secret" Facebook group where they can support one another in healthy lifestyle change. Finally, participants will have an opportunity to take part in a neighborhood tree planting campaign.
  Arms: Exploratory; RCT Intervention

SUMMARY:
The purpose of this study is to learn if a new whole-person lifestyle program improves the health of low-income mothers.

DETAILED DESCRIPTION:
This study will employ a randomized controlled trial (RCT) design to test a newly developed obesity reduction program, Koa Family, among overweight or obese mothers. An exploratory, uncontrolled study will assess its acceptance among normal-weight mothers.

Koa Family consists of a 6-month whole-person lifestyle program (WPLP) combined with text messaging and social media support and the opportunity to take part in a neighborhood tree planting campaign. This multi-pronged program is intended to reduce weight in the short-term while building self-empowerment and connections to community resources so that participants can sustain long-term weight loss.

Koa Family will be implemented in select communities in Yolo and Sacramento counties, California. Overweight or obese study participants will be randomized to either an intervention or control group; all normal-weight participants will be assigned to the intervention. All participants will complete a survey and have their height and weight measured at baseline and 3-, 6-, 9- and 12-month follow-up. Intervention participants will also take part in a focus group at the 3-month midpoint of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Comfortable speaking and reading English
* Primary caregiver for ≥1 child, aged 3-17, who lives at home
* Living in a low-income household (at or below 185% of the Federal Poverty Level)
* Living in the study site catchment area
* Ability to receive and send text messages
* BMI ≥ 25 kg/m2 for RCT study
* BMI ≥18.5 and <25 kg/m2 for exploratory study

Exclusion Criteria:

* Pregnant
* Breastfeeding
* Within 2 years postpartum
* Life-threatening illness
* Institutionalization (i.e., not free-living in the community)
* Moderate to severe mental illness
* Receiving nutrition therapy from a health or health care provider (licensed or unlicensed)
* Had or are considering bariatric surgery
* Medically diagnosed eating disorder
* Taking medication that affects weight
* Thyroid disease
* Type 1 or Type 2 diabetes without medical clearance from the participant's physician
* Plans to move away from study site catchment area during the one-year study period

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 149 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (kg/m2) | 12 months
  Objectively measured

SECONDARY OUTCOMES:
Change in diet quality | 12 months
  Fruit and vegetable consumption and other indicators calculated from 24-hour dietary recall
Change in physical activity | 12 months
  Self-report moderate-intensity equivalent minutes per week calculated from the BRFSS Physical Activity Rotating Core questionnaire
Change in health-related quality of life | 12 months
  Summary score from SF-36v2 instrument
Cost effectiveness | 12 months
  Dollars per change in BMI and quality-adjusted life-year (QALY)

CONTACTS AND LOCATIONS:
Overall Officials: Desiree R Backman, DrPH, MS, RD, Principal Investigator — UC Davis; Kenneth W Kizer, MD, MPH, Study Director — UC Davis
Locations (1):
- UC Davis Institute for Population Health Improvement, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No